CLINICAL TRIAL: NCT04872517
Title: Detecting Changes Before and After Chemotherapy or Radiotherapy in Patients With Head and Neck Cancer by Meridian Electroacupuncture Analysis Device (MEAD)
Brief Title: Meridian Energy Changes of Head and Neck Cancer Patients After Chemotherapy or Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liao Jian An (Other)
Responsible Party: Sponsor-Investigator, Liao Jian An, Attending physician of Traditional Chinese Medicine department, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202100209B0C501
Record Dates: First submitted 2021-04-27; First posted 2021-05-04 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: This research will use instruction named MEAD to detect the meridian energy before and after chemotherapy or/and radiotherapy. MEAD is a non-invasive device, it will not inter the conventional treatment that conduct by hematology oncology department and radiation oncology department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 34 head and neck cancer patients, expected to proceed chemotherapy or radiotherapy in hospital. (Experimental): Total 34 anticipants will recruit in this research. Age was limited between 20years old to 75 years old. All of anticipants agree to join this trail and be followed through treatment , and without underlying disease that threaten life.
  Interventions: Device: Meridian Electroacupuncture Analysis Device (MEAD)

INTERVENTIONS:
Device: Meridian Electroacupuncture Analysis Device (MEAD) — use MEAD to detect energy change in patient with head and neck cancer

SUMMARY:
This trial is conducted by using MEAD to detect the meridian changes in patients with head and neck cancer after conventional treatment of chemotherapy or radiotherapy.

DETAILED DESCRIPTION:
The purpose of this research is observe the change of meridian energy in patients have be diagnosed with head and neck cancer. The instrument we use is a non-invasive device called meridian energy analysis device(MEAD). The theory of MEAD is use conductive rod to measure the skin resistance from the specific point in human body, and to calculate the meridian's energy change. In Traditional Chinese Medicine theory, physician doctor believe that the median in human body would be affected by disease or uncomfortable condition. So, this time, we who a group of physician of Traditional Chinese medicine department conduct this research to assess the energy change in patients with head and neck cancer. The trail cooperate with radiation oncology department and hematology oncology department. Subject enrollment from radiation oncology department and hematology Oncology department. All of subjects have be diagnosed with head and neck cancer, and will to receive conventional treatment, no matter chemotherapy or/and radiotherapy.

The major assessment of our research is meridian energy by MEAD before treatment, and six consecutive cycles. In addition to this, pain degree, oral mucositis condition, impact on life quality, and blood test, diagnosis imaging data will be collected.

According to G*Power( 3.1.9.4 edition), we expected to recruit 34 subjects. All of Statistical Analysis will use SPSS, pair-t test is used to analyze continuous variable, categorical variable will be analyzed by Chi-Square Test. Multivariate regression analysis will be apply to discuss the major factor of the meridian changes.

MEAD is a kind of non-invasive device, hasn't had adverse effect until now. We will start emergency handling If accidents happened within measurement.

ELIGIBILITY:
Inclusion Criteria:

1. patients with head and neck cancer, included nasopharyngeal carcinoma, laryngeal cancer, oropharyngeal cancer, ear and oral cancer, hypopharyngeal cancer, salivary-gland carcinoma. Aged between 20 years old to 75years old, no gender difference.
2. patients with head and neck cancer has not received surgery yet, and will plan to accept chemotherapy and/or radiotherapy.
3. recurrent head and neck cancer, and expect to received chemotherapy and/or radiotherapy.
4. patient with vital sings stableness, conscious clear, and have ability to recognize the contain of trail and sign consent.
5. not accept other adjuvant therapy.
6. no brain metastasis or psychosis, and will to join whole course as well as accept assessments.

Exclusion Criteria:

1. Aged less than 20 years old and over 75 years old。
2. Patients be diagnosed with head and neck cancer, and accepted surgery, or already finished chemotherapy and/or radiotherapy.
3. patient with brain metastasis, conscious unclear, and have not able to recognize the contain of trail and sign consent.
4. Accept other adjuvant therapy and chemotherapy and/or radiotherapy simultaneously.
5. Combined with serious organs failure。
6. Have contraindication in chemotherapy or radiotherapy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
meridian energy | An average of 6 weeks
  energy change in meridian

SECONDARY OUTCOMES:
the number of participants with blood test data abnormal | An average of 6 weeks
  calculate the ratio of participants in hemodynamic alteration whom accept chemotherapy or/and radiotherapy, and compare the hemodynamic change with meridian energy change. Blood test include CBC/DC (WBC, RBC, Hemoglobin, Hematocrit, platelets, segment, lymphocyte, absolutely neutrophil), GOT/GPT, Bun/Creatinine, Bilirubin.
pain degree | An average of 6 weeks
  use Numerical Rating Scale(0-10) to assess.
Oral mucositis grading | An average of 6 weeks
  compare enrollment subjects's oral condition with picture from MASCC/ISOO clinical practice guidelines (grade 0-grade 4)
adverse impact on quality of life | An average of 6 weeks
  use EORTC QLQ - H&N35 questionnaire to evaluate the treatment impact on subject feeling
imaging diagnosis | An average of 6 weeks
  compare tumor condition in diagnostic image data (shrink or progress) with the energy change in meridian.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-An Liao, Principal Investigator — medical attending
Locations (1):
- Chang Cung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No